CLINICAL TRIAL: NCT00854516
Title: Open Label Clinical Study to Assess the Clinical Safety of a New Compression Procedure in Subjects With Peripheral Arterial Vascular Disease
Brief Title: Open Label Clinical Study to Assess the Clinical Safety of a New Compression Device in Subjects With Peripheral Arterial Vascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU Study No-05-000007
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Arterial Vascular Disease
Keywords: compression therapy; 3M
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: A new treatment approach is to have an effective working pressure combined with a low resting pressure. — Procedure Schedule: The total duration for study participation will be 14 days (8 visits).
  Subject eligibility will be determined at the initiation visit. All eligible subjects will receive the compression device on the study leg and will return to the clinical center at day 1, 2, 3, 4, 7, 10 and 14 to assess safety. At each clinical visit (except visit day 14) the compression device will be reapplied. The study participation ends after 14 days.

SUMMARY:
To assess the safety of a new compression device applied to patients with an ankle brachial pressure index (ABPI) 0,5 - 0,8 who are treated for two weeks in daily routine practice. Several perfusion assessments will investigate safety under reduced compression therapy.

DETAILED DESCRIPTION:
Venous leg ulcers represent a very common clinical problem with increasing prevalence in an aging population. It is believed that venous insufficiency is the underlying condition responsible for 54-81% of leg ulcers. About 8% of leg ulcers are related to arterial insufficiency and about 14% have a mixed aetiology. Compression therapy is considered the most effective treatment for these ulcers. The overall cost of chronic venous leg ulcer is high because long term ongoing care is required. Also the quality of life of these patients is jeopardized due to long lasting ulcer treatments and inconvenient compression therapies.

Several compression products are available on the market and there is a large body of literature describing the clinical benefit of different compression systems.

A new treatment approach with the new device is to have an effective working pressure combined with a low resting pressure. A high working pressure achieved by a rigid sleeve around a patient's leg is essential to support the muscle pump, necessary for sufficient blood reflux. However the resting pressure could be low without relevant reduction of compression efficacy but with an increase in safety for patients with a mild to moderate peripheral arterial occlusive disease (PAOD). A high resting pressure is believed to be a main reason for reduced arterial skin perfusion which can result in pressure related skin damage. Accordingly most compression systems are not indicated for patients with an ABPI lower than 0.8. About 25% of patients with chronic venous insufficiency suffer from PAOD and hence are very difficult to treat with compression. With the new device, these patients could be sufficiently treated, because a low resting pressure is believed to have low influence on skin perfusion.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age 18 years or older.
2. Subjects suffering from peripheral arterial occlusive disease (PAOD) with an ABPI (ankle brachial pressure index) of the treated leg between 0.5 - 0.8 as measured within up to 4 weeks prior to enrollment. About 5 subjects of the study population should have an ABPI of 0.5.
3. Subjects who are co-operative, willing to give written informed consent prior to study entry and willing to comply with the study protocol.
4. Subjects who can walk (with or without a walking aid).

   -

Exclusion Criteria:

1. Subjects with an ABPI < 0.5 or > 0.8 as measured within up to 4 weeks prior to enrollment.
2. Subjects whose general condition, in the opinion of the investigator, preclude for compression therapy.
3. Subjects with paralysis of the study leg
4. Subjects who started or significantly changed treatment with mood altering substances (e.g. antidepressant drugs) within two weeks prior to enrollment.
5. Subjects with significant instable coagulopathy; subjects treated with anticoagulant therapeutics can be included.
6. Subjects who are participating in any prospective clinical study that can potentially interfere with this study.
7. Subjects who are, in the opinion of the clinical investigator, unsuitable for enrollment in this study, for reasons not specified in the exclusion criteria.
8. Subjects with known allergies to other materials in the compression device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the safety of the new compression device in subjects with an ankle brachial pressure index (ABPI) between 0.5-0.8. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Juenger, Prof. Dr. MD, Principal Investigator — Universitaetsklinikum Greifswald
Locations (1):
- Universitaetsklinikum Greifswald, Greifswald, Germany